CLINICAL TRIAL: NCT03734757
Title: Interest of Trimodality PET-CT Choline MRI Before Radiotherapy in High Risk Prostate Cancer Using Geometric Indexes
Brief Title: Interest of Trimodality PET-CT Choline MRI Before Radiotherapy in High Risk Prostate Cancer
Acronym: DEMETER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB18.02
Record Dates: First submitted 2018-10-31; First posted 2018-11-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; Imaging; trimodality
MeSH Terms: conditions — Prostatic Neoplasms | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trimodality (Experimental): PET-CT with fluorocholine and MRI
  Interventions: Procedure: imaging in trimodality

INTERVENTIONS:
Procedure: imaging in trimodality — PET-CT and MRI

SUMMARY:
The initial staging of locally advanced prostate cancer is made with Computed Tomography scan (CT), Magnetic Resonance Imaging (MRI), and bone scan (BS).

For this type of cancer, reference treatment is radiotherapy combined with hormone therapy.

The added value of MRI in the delineation of volumes for radiotherapy is known, especially for the definition of extra-prostatic extensions and prostatic apex. However, its regular use is difficult. Indeed, acquisition of Magnetic Resonance Imaging parameters for diagnostic are not adapted to be fused with the planning Computed Tomography.

The literature shows that Positron Emission Tomography-Computed Tomography with Fluorocholine is better in terms of diagnostic performance compared to bone scan for bone metastases and to pelvic Magnetic Resonance Imaging for nodal extension.

It would therefore improve staging for these patients with a high risk of locoregional and metastatic invasion even if its use is currently not recommended in the initial staging.

Thanks to Magnetic Resonance Imaging acquisition parameters adapted to Radiotherapy and additional functional information, an acquisition in tri-modality Positron Emission Tomography/computed Tomography/ Magnetic Resonance Imaging could have an impact on the volumes definition for radiotherapy or even on the therapeutic strategy.

The aim of the study is to evaluate the volume modifications obtained on the trimodality evaluation, compared to the standard initial staging (geometric comparison).

In addition, it would be a preliminary study for a project using Prostate-specific membrane antigen (PSMA) in trimodality, and / or for a therapeutic interventional study.

DETAILED DESCRIPTION:
Prostate cancer (Pca) is the first human cancer in terms of incidence and the third leading cause of tumor death (56,000 new cases/year in France in 2012 and nearly 9,000 deaths). According to the French Association of Urology 2013, an individual screening based on rectal examination and prostatic specific antigen (PSA) is recommended for men over 50. Ultrasound (US) guided biopsy allows the histological diagnosis and the Gleason score evaluation. For high-risk of prostate Cancer, initial staging is based on pelvic Magnetic Resonance Imaging, abdominal pelvic computed tomography and bone scan.

External radiotherapy combined with prolonged hormone therapy is the reference treatment for these cancers.

Radiotherapy requires a planning Computed Tomography. Magnetic Resonance Imaging is known to be better for definition of extra-prostatic extensions and prostatic apex. However, its regular use is difficult for the radiotherapy planning.

Moreover, Positron Emission Tomography-Computed Tomography with Fluorocholine detects earlier nodal and bone metastasis.

Hypothesis: A single planning acquisition in trimodality in radiotherapy position should improve simultaneously the initial staging and the volume delineation for radiotherapy.

Main objective: Main objective is to compare volumes delineation (prostatic target and organ at risk) thanks to geometric index (Jaccard, Dice and overlap), got by trimodality and by standard initial staging and planning Computed Tomography.

Expected results: Thanks to literature data, it can be expected that prostatic delineation target volume will significantly decrease with Magnetic Resonance Imaging.

Furthermore, thanks to Positron Emission Tomography-Computed Tomography with Fluorocholine, radiotherapy planning would be different, detecting 14% of nodal extension and 7% of bone metastasis.

Finally, with trimodality the investigators expect a smaller prostate volume and a higher detection of metastatic lymph node or bone metastasis.

Then, the investigators expect an improvement of the management of patients by:

* Detecting more nodal or bone metastasis and avoiding a useless local treatment by radiotherapy
* Improving prostatic target volume delineation and allowing a better protection of organ at risk.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years
* prostate cancer : High risk (according to D'Amico Classification)
* and/or Node positive on MRI
* T2c-T3 on MRI
* with staging assessment
* will receive radiotherapy

Exclusion Criteria:

* second cancer
* contraindication to MRI
* participation in an another therapeutic trial
* patients under guardianship or curatorship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Delineation volumes | 1 day
  Measure of volumes delineation for radiotherapy thanks to trimodality and comparison to those obtained with standard technique

SECONDARY OUTCOMES:
Treatment plan | 6 weeks
  percentage of patient for whom the therapeutic decision will be different with standard assessment
Dosimetry | 6 weeks
  Variation of dosimetry between trimodality imaging and standard assessment
F-choline fixation in MRI | 1 day
  Comparison of percentage of choline fixation during magnetic resonance imaging
contouring of target lesions and organ at risk | 6 weeks
  comparison of contouring duration with the two techniques of imagery

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No